CLINICAL TRIAL: NCT02849626
Title: An Open-Label, Multicenter Study With an Extension Phase to Evaluate the Safety, Tolerability, and Exposure-Efficacy Relationship of Perampanel Oral Suspension When Administered as an Adjunctive Therapy in Pediatric Subjects (Age 4 to Less Than 12 Years) With Inadequately Controlled Partial-Onset Seizures or Primary Generalized Tonic Clonic Seizures
Brief Title: Perampanel as Adjunctive Therapy in Pediatrics With Partial Onset Seizures or Primary Generalized Tonic Clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-311; 2014-002167-16 (EudraCT Number)
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Partial-Onset or Primary Generalized Tonic-Clonic Seizures
Keywords: Partial-Onset Seizures; Primary Generalized Tonic-Clonic Seizures; Adjunctive Therapy; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perampanel (Experimental): Perampanel 0.5 milligrams per milliliter (mg/mL) oral suspension
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — E2007

SUMMARY:
This is an open-label, multicenter study with an Extension Phase to evaluate the safety and tolerability of perampanel oral suspension when administered as an adjunctive therapy in children (ages 4 to less than [<] 12 years) with inadequately controlled partial onset seizures (POS) or primary generalized tonic clonic (PGTC) seizures.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm study in children (age 4 to <12 years) with inadequately controlled POS or PGTC seizures. The study will consist of a Core Phase and two Extension Phases (Extension Phase A [for all countries in the study], and Extension Phase B [available for participants enrolled in Japan and in countries where an extended access program {EAP} cannot be implemented, after completion of Extension Phase A]). The Core Phase will consist of the following 2 phases: Pretreatment and Treatment Phase. The Pretreatment Phase, during which participants will be assessed for eligibility, will consist of up to a 4-weeks +/- 3 days Screening/Baseline Period. The Treatment Phase will consist of 3 periods: Titration Period (up to an 11-weeks: dose titration on the basis of individual clinical response and tolerability), Maintenance Period (up to a 12-weeks: continuation of perampanel oral suspension once daily at the dose level achieved at the end of the Titration Period), and Follow-up Period (up to 4-weeks +/- 7 days: only for those participants not entering into Extension Phase A or those who prematurely discontinue from the study). Extension Phase A will consist of up to 29-weeks Maintenance Period and up to 4-weeks +/- 7 days Follow-up Period after the last dose of perampanel only for participants who did not enter into Extension Phase B. All participants who complete all scheduled visits up to and including Visit 9 in the Treatment Phase will be eligible to participate in Extension Phase A of the study. During the Maintenance Period of Extension Phase A, all participants will continue with their optimal perampanel dose (that is, dose level that they complete on during the Core Phase). After completing Extension Phase A, participants in Japan and in countries where EAP cannot be implemented, participants will be eligible to participate in Extension Phase B. In Japan, treatment will continue as long as clinically appropriate according to the judgment of the investigator. However, treatment of participants in Extension B will be completed when the participant reaches 12 years of age or when perampanel is commercially available in Japan for treatment of POS in pediatric participants (4 to less than 12 years of age). In countries where an EAP cannot be implemented, participation in Extension B will continue as long as clinically appropriate according to the judgment of the investigator, until the participants reaches 12 years of age or perampanel oral suspension is commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of epilepsy with POS with or without secondarily generalized (SG) seizures or PGTC seizures according to the International League Against Epilepsy's (ILAE) Classification of Epileptic Seizures (1981). A diagnosis should have been established at least 6 months prior to Visit 1 by clinical history and an electroencephalogram (EEG) that is consistent with the diagnosis; normal interictal EEGs will be allowed provided that the participant meets the other diagnosis criterion (that is, clinical history)
* Male or female participant, from age 4 to <12 years at the time of informed consent/assent
* Have a minimum weight of 16 kilograms (kg) (35 pounds [lb])
* Have had a brain imaging (example, magnetic resonance imaging [MRI] scan or computed tomography [CT] before Visit 1 that ruled out a progressive cause of epilepsy)
* During the 12 weeks +/- 3 days (4 weeks +/- 3 days in Japan only) prior to Visit 2, participants must have equal or greater than (=>) one POS or one PGTC seizure. Only simple POS with motor signs, complex POS, and complex POS with secondary generalization are counted toward this inclusion for POS
* Are currently being treated with stable doses of 1 to a maximum of 3 approved antiepileptic drugs (AEDs). Doses must be stable for at least 4 weeks before to Visit 1; in the case where a new AED regimen has been initiated for a participant, the dose must be stable for at least 8 weeks prior to Visit 1. Only one EIAED (defined as carbamazepine, phenytoin, oxcarbazepine, or eslicarbazepine) out of the maximum of three AEDs is allowed (A vagal nerve stimulator [VNS] will be counted as one of the 3 allowed AEDs)

Exclusion Criteria:

* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta human chorionic gonadotropin [β-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 International Units per liter [IU/L] or equivalent units of β-hCG or hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (example, total abstinence, an intrauterine device, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation. If a highly effective method is not appropriate or acceptable for the participant, then the participant may use a medically effective method (example, a double barrier method such as condom plus diaphragm with spermicide)
  * Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from being sexually active during the study period or for 28 days after study drug discontinuation
  * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation
* Current or history of pseudo-seizures (psychogenic nonepileptic seizures) within approximately 5 years before Visit 1
* Have a history of status epilepticus that required hospitalization during the 6 months before Visit 1
* Have an unstable psychiatric diagnosis that may confound participants' ability to participate in the study or that may prevent completion of the protocol-specified tests (example, significant suicide risk, including suicidal behavior and ideation within 6 months before Visit 1, current psychotic disorder, acute mania)
* Any suicidal ideation with intent with or without a plan within 6 months before Visit 2 (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale [C-SSRS]) in participants aged 6 and above
* Are scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1; however, those who have previously documented "failed" epilepsy surgery will be allowed
* Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Evidence of moderate or severe renal insufficiency as defined by estimated glomerular filtration rates (eGFRs) of 31 to <60 milliliters per minute (mL/min) and <30 mL/min, respectively
* Evidence of significant active hepatic disease. Stable elevation of liver enzymes, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) due to concomitant medication(s), will be allowed if they are less than 3 times the upper limit of normal (ULN)
* Evidence of significant active hematological disease; white blood cell (WBC) count equal or less than (=<) 2500 per (/) microliter (µL) (2.50 1 constant [E]+09/liter [L]) or an absolute neutrophil count =<1000/µL (1.00 1E+09/L)
* Clinically significant electrocardiogram (ECG) abnormality, including prolonged corrected QT interval (QTc) defined as greater than (>) 450 milliseconds (msec)
* Have a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors
* Multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (example, Stevens Johnson syndrome), hematological, or organ toxicity reactions.
* Concomitant use of felbamate as an AED for <2 years or where the dose has not been stable for at least 8 weeks before Visit 1. Participants must not have a history of WBC count =<2500/µL, platelets below 100,000, liver function tests (LFTs) above 3 times the ULN, or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If participants received felbamate in the past, it must have been discontinued 8 weeks before Visit 1 to be eligible for study participation
* Concomitant use of vigabatrin: participants who took vigabatrin in the past must be off vigabatrin for at least 5 months before Visit 1 and with documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in a visual perimetry test
* Concomitant use of cannabinoids
* Used benzodiazepines for epilepsy during which the dose has not been stable for >4 weeks prior to Visit 1. Benzodiazepines use as rescue medication for seizure control is allowed; however, intermittent use of benzodiazepines for any other indication (example, anxiety/sleep disorders) is prohibited
* A VNS implanted <5 months before Visit 1 or changes in parameter <4 weeks before Visit 1 (or thereafter during the study)
* On a ketogenic diet for which the diet is not a stable regimen for at least 4 weeks before Visit 1
* History of or a concomitant medical condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study or compromise the participant's ability to safely complete the study
* Have previously been exposed to perampanel in a clinical trial or by prescription for more than 2 months or discontinued for Adverse Events (AEs)
* Have participated in a study involving administration of an investigational drug or device within 4 weeks before Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer
* Participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Information — Eisai Inc.
Locations (91):
- United States (29):
  - Facility #1, Little Rock, Arkansas
  - Facility #1, Palo Alto, California
  - Facility #1, Aurora, Colorado
  - Facility #1, Gulf Breeze, Florida
  - Facility #1, Loxahatchee Groves, Florida
  - Facility #1, Orlando, Florida
  - Facility #1, Atlanta, Georgia
  - Facility #1, Savannah, Georgia
  - Facility #1, Boise, Idaho
  - Facility #1, Chicago, Illinois
  - Facility #1, Urbana, Illinois
  - Facility #1, Ames, Iowa
  - Facility #1, Wichita, Kansas
  - Facility #1, Lexington, Kentucky
  - Facility #2, Lexington, Kentucky
  - Facility #1, New Orleans, Louisiana
  - Facility #1, Duluth, Minnesota
  - Facility #1, Kansas City, Missouri
  - Facility #1, Henderson, Nevada
  - Facility #1, Hackensack, New Jersey
  - Facility #1, Voorhees Township, New Jersey
  - Facility #1, Brooklyn, New York
  - Facility #1, Winston-Salem, North Carolina
  - Facility #1, Cleveland, Ohio
  - Facility #1, Memphis, Tennessee
  - Facility #1, Austin, Texas
  - Facility #1, San Antonio, Texas
  - Facility #1, Tacoma, Washington
  - Facility #1, Milwaukee, Wisconsin
- Belgium (5):
  - Facility #1, Pulderbos, Antwerpen
  - Facility #1, Ottignies, Brabant Wallon
  - Facility #1, Brussels, Brussels Capital
  - Facility #1, La Louvière, Hainaut
  - Facility #1, Brussels
- Canada (2):
  - Facility #1, Calgary, Alberta
  - Facility #1, Montreal, Quebec
- Czechia (2):
  - Facility #1, Ostrava
  - Facility #1, Prague
- France (7):
  - Facility #1, Marseille, Bouches-du-Rhone
  - Facility #1, Lille
  - Facility #1, Marseille
  - Facility #1, Paris
  - Facility #2, Paris
  - Facility #1, Strasbourg
  - Facility #1, Toulouse
- Hungary (4):
  - Facility #1, Budapest
  - Facility #2, Budapest
  - Facility #1, Miskolc
  - Facility #1, Pécs
- Italy (5):
  - Facility #1, Mantova, Lombardy
  - Facility #1, Calambrone, Tuscany
  - Facility #1, Bologna
  - Facility #1, Florence
  - Facility #1, Milan
- Japan (22):
  - Eisai Trial Site #1, Sapporo, Hokkaido
  - Eisai Trial Site #1, Zentsujichó, Kagawa-ken
  - Eisai Trial Site #1, Sendai, Miyagi
  - Eisai Trial Site #1, Hamamatsu, Shizuoka
  - Eisai Trial Site #1, Fukuoka
  - Eisai Trial Site #1, Gifu
  - Eisai Trial Site #1, Hakodate-shi
  - Eisai Trial Site #1, Hiroshima
  - Eisai Trial Site #1, Izumi
  - Eisai Trial Site #1, Kobe
  - Eisai Trial Site #1, Kumamoto
  - Eisai Trial Site #1, Nagoya
  - Eisai Trial Site #1, Nara
  - Eisai Trial Site #1, Niigata
  - Eisai Trial Site #1, Okayama
  - Eisai Trial Site #1, Osaka
  - Eisai Trial Site #1, Ōmura
  - Eisai Trial Site #1, Sagamihara
  - Eisai Trial Site #1, Sapporo
  - Eisai Trial Site #1, Shizuoka
  - Eisai Trial Site #1, Yamagata
  - Eisai Trial Site #1, Yokohama
- Facility #1, Riga, Latvia
- Poland (3):
  - Facility #1, Poznan, Greater Poland Voivodeship
  - Facility #1, Gdansk, Pomeranian Voivodeship
  - Facility #1, Kielce, Świętokrzyskie Voivodeship
- South Korea (5):
  - Facility #1, Daegu
  - Facility #1, Daejeon
  - Facility #1, Seoul
  - Facility #2, Seoul
  - Facility #3, Seoul
- Spain (6):
  - Facility #1, Esplugues de Llobregat, Barcelona
  - Facility #1, Barcelona
  - Facility #2, Barcelona
  - Facility #1, Madrid
  - Facility #1, Seville
  - Facility #1, Valencia

REFERENCES:
- [Derived] Trigg A, Brohan E, Cocks K, Jones A, Tahami Monfared AA, Chabot I, Meier G, Campbell R, Li H, Ngo LY. Health-related quality of life in pediatric patients with partial onset seizures or primary generalized tonic-clonic seizures receiving adjunctive perampanel. Epilepsy Behav. 2021 May;118:107938. doi: 10.1016/j.yebeh.2021.107938. Epub 2021 Apr 8. PMID 33839450
- [Derived] Fogarasi A, Flamini R, Milh M, Phillips S, Yoshitomi S, Patten A, Takase T, Laurenza A, Ngo LY. Open-label study to investigate the safety and efficacy of adjunctive perampanel in pediatric patients (4 to <12 years) with inadequately controlled focal seizures or generalized tonic-clonic seizures. Epilepsia. 2020 Jan;61(1):125-137. doi: 10.1111/epi.16413. Epub 2020 Jan 7. PMID 31912493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 58 investigative sites in the United States, European Union and Asia Pacific from 16 November 2016 to 06 December 2021.
Pre-assignment Details: A total of 208 participants were screened; of which 28 were screen failures; 180 received study treatment in Core Phase. Of 146 participants who completed the Core Phase, 136 entered Extension Phase A. Of 122 who completed Extension Phase A, 42 received treatment in Extension B. Study has a Core Phase and two Extension Phases (Phase A and Phase B). In Extension Phase B only safety data was collected for participants who could not enroll in an extended access program (EAP).
Groups:
- Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS: Core Phase: Participants with partial onset-seizures (POS) received perampanel 0.5 milligrams per milliliter (mg/mL) oral suspension titrated beyond 8 milligram per day (mg/day) up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any enzyme-inducing antiepileptic drug [EIAED]), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel once daily at optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed Core Phase, entered Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
- Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures: Core Phase: Participants with primary generalized tonic clonic (PGTC) seizures received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any other EIAED), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel oral suspension once daily at the optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed the Core Phase, entered the Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
- Extension B: Perampanel 0.5 mg/mL: POS; Extension B: Perampanel 0.5 mg/mL: PGTC Seizures: Participants who completed Core Phase and Extension Phase A and eligible for Extension Phase B entered Extension Phase B, and continued with their optimal perampanel dose from Core Phase until a participant reached 12 years of age, switched to the commercial perampanel product, or discontinued for safety or administrative reasons.
Period: Core Phase (up to 23 Weeks)
Arm/Group | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures | Extension B: Perampanel 0.5 mg/mL: POS | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures
Started | 149 | 31 | 0 | 0
Completed | 122 | 24 | 0 | 0
Not Completed | 27 | 7 | 0 | 0
Not completed — Adverse Event | 11 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 0 | 0
Not completed — Inadequate Therapeutic Effect | 6 | 2 | 0 | 0
Not completed — Non-specified | 3 | 0 | 0 | 0
Period: Extension Phase A (up to 29 Weeks)
Arm/Group | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures | Extension B: Perampanel 0.5 mg/mL: POS | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures
Started | 116 (Only eligible participants who completed Core Phase entered into Extension Phase A.) | 20 (Only eligible participants who completed Core Phase entered into Extension Phase A.) | 0 | 0
Completed | 105 | 17 | 0 | 0
Not Completed | 11 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Inadequate Therapeutic Effect | 3 | 1 | 0 | 0
Not completed — Non-specified | 1 | 0 | 0 | 0
Period: Extension Phase B (up to 89 Weeks)
Arm/Group | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures | Extension B: Perampanel 0.5 mg/mL: POS | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures
Started | 0 | 0 | 41 (Participants who completed Core and Extension Phase A and could not enroll into EAP entered into Extension Phase B.) | 1 (Participants who completed Core and Extension Phase A and could not enroll into EAP entered into Extension Phase B.)
Completed | 0 | 0 | 36 | 1
Not Completed | 0 | 0 | 5 | 0
Not completed — Inadequate Therapeutic Effect | 0 | 0 | 3 | 0
Not completed — Participant choice | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Groups:
- Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS: Core Phase: Participants with partial onset-seizures (POS) received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any EIAED, or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel once daily at optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed Core Phase, entered Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures | Total
Number analyzed (Participants) | 149 | 31 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (2.10) | 8.5 (2.03) | 8.1 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 11 | 88
  Male | 72 | 20 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 141 | 19 | 160
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 23 | 93
  Black or African American | 2 | 1 | 3
  Japanese | 65 | 0 | 65
  Other Asian | 5 | 1 | 6
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 2 | 1 | 3
  Missing | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs) for Total Group of Participants - Core Phase and Extension Phase A of This Study
Time Frame: Baseline up to 4 weeks (follow up in Extension Phase A) after last dose of study drug in Extension Phase A at Week 52 (up to 56 weeks)
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: percentage of participants
Groups:
- Perampanel 0.5 mg/mL: All Participants: Core Phase: Participants with POS or PGTC seizures received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any EIAED), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel once daily at optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed Core Phase, entered Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 180
percentage of participants
  Treatment Emergent AEs | 90.0
  Treatment Emergent SAEs | 20.0

2. Primary Outcome: Percentage of Participants With Treatment Emergent Markedly Abnormal Laboratory Values for Total Group of Participants- Core Phase and Extension Phase A of This Study
Time Frame: Baseline up to 52 weeks
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure and number analyzed 'n' signifies participants who were evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 177
percentage of participants
  Potassium: Markedly Abnormal High | 0.6
  Sodium: Markedly Abnormal Low | 1.1
  Alanine Aminotransferase: Abnormal High | 1.1
  Calcium: Abnormal Low | 0.6
  Gamma Glutamyl Transferase: Abnormal High | 2.8
  Neutrophils: Abnormal Low: number analyzed (Participants) | 176
  Neutrophils: Abnormal Low | 9.1
  Hemoglobin: Abnormal Low: number analyzed (Participants) | 176
  Hemoglobin: Abnormal Low | 1.7
  Leukocytes: Abnormal Low: number analyzed (Participants) | 176
  Leukocytes: Abnormal Low | 0.6

3. Primary Outcome: Percentage of Participants With Abnormal Vital Sign Values for Total Group of Participants- Core Phase and Extension Phase A of This Study
Description: Pre-defined criteria of vital signs abnormalities: maximum (max.) increase or decrease from baseline in sitting/supine systolic blood pressure (SBP) of greater than or equal to (>=) 20 or 40 millimeter of mercury (mmHg); maximum increase or decrease from baseline in sitting/supine diastolic blood pressure (DBP) >=10 or 20 mmHg; increase or decrease from baseline in pulse rate (number of heart beats per minute [bpm]) of >=15 or 30 bpm. Data for this outcome measure has been assessed and reported till Week 52.
Time Frame: Baseline up to 52 weeks
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 179
percentage of participants
  Systolic Blood Pressure: Increment >=20 mmHg | 24.6
  Systolic Blood Pressure: Increment >=40 mmHg | 2.2
  Systolic Blood Pressure: Decrement >=20 mmHg | 20.1
  Systolic Blood Pressure: Decrement >=40 mmHg | 0.6
  Diastolic Blood Pressure: Increment >=10 mmHg | 48.0
  Diastolic Blood Pressure: Increment >=20 mmHg | 26.8
  Diastolic Blood Pressure: Decrement >=10 mmHg | 38.0
  Diastolic Blood Pressure: Decrement >=20 mmHg | 16.8
  Pulse: Increment >=15 bpm | 35.8
  Pulse: Increment >=30 bpm | 11.7
  Pulse: Decrement >=15 bpm | 39.7
  Pulse: Decrement >=30 bpm | 13.4

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Electrocardiogram (ECG) Parameters for Total Group of Participants- Core Phase and Extension Phase A of This Study
Time Frame: Baseline up to 52 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 174
percentage of participants
  QTc Bazett: Increase of >30 millisecond (msec) | 8.0
  QTc Bazett: Increase of >60 msec | 0
  QTc Bazett: >450 msec | 4.0
  QTc Bazett: >480 msec | 0
  QTc Bazett: >500 msec | 0
  QTc Fridericia: Increase of >30 msec | 5.2
  QTc Fridericia: Increase of >60 msec | 0
  QTc Fridericia: >450 msec | 0
  QTc Fridericia: >480 msec | 0
  QTc Fridericia: >500 msec | 0

5. Secondary Outcome: Model Predicted Percent Change in Average Seizure Frequency Over 28 Days During Maintenance Period in Core Phase of This Study From Baseline- Assessed as Relationship With Average Steady State Plasma Concentration (Cav, ss) of Perampanel (518 ng/mL)
Description: Seizure frequency derived from information (seizure count and type) recorded in participant diary. Seizure frequency per 28 days was calculated as number of seizures divided by number of days in interval; multiplied by 28. Due to sparse pharmacokinetic (PK) sampling in study, data of endpoint was analyzed by pooling data from other Phase II and III studies of perampanel along with data of this current study, including participants with POS or PGTC. Only data for participants taking perampanel 8 mg/day (corresponding to Cav, ss of 518 ng/mL) were reported. Participants taking perampanel 12 mg/day in studies from which data were pooled, were not included in analysis for this measure. Here, ng/mL= nanogram per milliliter. Data for this measure was calculated through model prediction; reported as "percent change" with measure type as "number" and measure dispersion as "Not applicable, NA".
Time Frame: Baseline, Week 23
Population: All participants who received perampanel who have seizure frequency, cognition, or AE data with documented dosing history. Population for this measure included participants from other studies as well participants from this current study. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percent change
Groups:
- Perampanel: POS: All participants with POS who received perampanel 0.5 mg/mL oral suspension (for participants with age less than [<] 12 years) or tablets (for participants with age >=12 years) titrated to a dose of up to 8 mg/day for up to 23 weeks in studies E2007-G000-304 (NCT00699972), E2007-G000-305 (NCT00699582), E2007-G000-306 (NCT00700310), E2007-J000-335 (NCT01618695) and this current study (E2007-G000-311).
- Perampanel: PGTC Seizures: All participants with PGTC seizures who received perampanel 0.5 mg/mL oral suspension (for participants with age <12 years) or tablets (for participants with age >=12 years) titrated to a dose of up to 8 mg/day for up to 23 weeks in studies E2007-G000-232 (NCT01527006) and E2007-G000-332 (NCT01393743) and this current study (E2007-G000-311).
Arm/Group | Perampanel: POS | Perampanel: PGTC Seizures
Number analyzed (Participants) | 1371 | 92
percent change | -43.1 | -63.6

6. Secondary Outcome: Overall Responder Probability For Non-Asian Participants With POS During Core Phase of This Study: Assessment Based on Relationship With Average Steady State Plasma Concentration (Cav, ss) of Perampanel
Description: For this outcome measure, responders were those who experienced a 50 percent (%) or greater reduction in seizure frequency per 28 days from baseline. Due to the sparse PK sampling in this study, the data of this outcome measure were pooled with data from other Phase III studies of perampanel conducted in participants with POS. "AEDs not affecting PK" refers to AEDs not affecting PK of perampanel. Data for this outcome measure has been reported for only non-Asian participants with POS per age groups. Responder probability has been reported for Cav,ss of perampanel when given along with different antiepileptic drugs (AEDs).
Time Frame: Baseline up to 23 weeks
Population: as for outcome 5
Measure: Number; unit: Responder probability
Groups:
- Perampanel: Participants Aged (<12 Years): All non-Asian participants with POS, received perampanel oral suspension (participants with age <12 years) titrated to a dose of up to 8 mg/day or up to 12 mg/day for up to 23 weeks in this current study E2007-G000-311.
- Perampanel: Participants Aged (>=12 Years): All non-Asian participants with POS, received perampanel tablets (participants with age >=12 years) titrated to a dose of up to 8 mg/day or up to 12 mg/day for up to 23 weeks in studies E2007-G000-304 (NCT00699972), E2007-G000-305 (NCT00699582), E2007-G000-306 (NCT00700310), E2007-J000-335 (NCT01618695).
Arm/Group | Perampanel: Participants Aged (<12 Years) | Perampanel: Participants Aged (>=12 Years)
Number analyzed (Participants) | 123 | 1420
Responder probability
  8 mg/day+ AEDs not affecting PK:Cav ss 518 ng/mL | 0.605 | 0.466
  12 mg/day+ AEDs not affecting PK:Cav ss 778 ng/mL | 0.669 | 0.535
  8 mg/day+ Oxcarbazepine/Phenytoin:Cav ss 258 ng/mL | 0.520 | 0.382
  12 mg/day+Oxcarbazepine/Phenytoin:Cav ss 387 ng/mL | 0.565 | 0.426
  8 mg/day+ Carbamazepine:Cav ss 175 ng/mL | 0.485 | 0.350
  12 mg/day+ Carbamazepine:Cav ss 263 ng/mL | 0.522 | 0.384

7. Secondary Outcome: Overall Responder Probability For Participants With PGTC Seizures During Core Phase of This Study: Assessment Based on Relationship With Average Steady State Plasma Concentration (Cav, ss) of Perampanel
Description: For this outcome measure, responders were those who experienced a 50% or greater reduction in seizure frequency per 28 days from baseline. Due to the sparse PK sampling in this study, the data of this outcome measure were analyzed by pooling the data from other Phase II and III studies of perampanel along with data of this current study, including participants with PGTC seizures. In this outcome measure, responder probability at different concentration values of perampanel when given with or without topiramate (an antiepileptic) has been reported.
Time Frame: Baseline up to 23 weeks
Population: as for outcome 5
Measure: Number; unit: Responder probability
Groups:
- Perampanel: Without Topiramate: All participants with PGTC seizures received perampanel as oral suspension (aged <12 years) or as oral tablets (aged >=12 years) titrated to a dose of up to 8 mg/day or up to 12 mg/day without topiramate for up to 23 weeks in studies E2007-G000-232 (NCT01527006) and E2007-G000-332 (NCT01393743) and this current study (E2007-G000-311).
- Perampanel: With Topiramate: All participants with PGTC seizures received perampanel as oral suspension (aged <12 years) or as oral tablets (aged >=12 years) titrated to a dose of up to 8 mg/day or up to 12 mg/day along with topiramate for up to 23 weeks in studies E2007-G000-232 (NCT01527006) and E2007-G000-332 (NCT01393743) and this current study (E2007-G000-311).
Arm/Group | Perampanel: Without Topiramate | Perampanel: With Topiramate
Number analyzed (Participants) | 138 | 31
Responder probability
  0 ng/mL | 0.46 | 0.26
  100 ng/mL | 0.71 | 0.50
  200 ng/mL | 0.74 | 0.54
  300 ng/mL | 0.76 | 0.57
  400 ng/mL | 0.77 | 0.58
  500 ng/mL | 0.78 | 0.59
  600 ng/mL | 0.79 | 0.60
  700 ng/mL | 0.80 | 0.61
  800 ng/mL | 0.80 | 0.62
  900 ng/mL | 0.80 | 0.63
  1000 ng/mL | 0.81 | 0.63
  1200 ng/mL | 0.82 | 0.64
  1400 ng/mL | 0.82 | 0.65
  1600 ng/mL | 0.82 | 0.66
  1800 ng/mL | 0.83 | 0.66
  2000 ng/mL | 0.83 | 0.67
  2200 ng/mL | 0.84 | 0.67
  2400 ng/mL | 0.84 | 0.68

8. Secondary Outcome: Number of Seizure Free Observations During Core Phase of This Study: Assessment Based on Relationship With Average Steady State Plasma Concentration (Cav, ss) of Perampanel
Description: Due to the sparse PK sampling in this study, the data of this outcome measure were analyzed by pooling data from other Phase II and III studies of perampanel along with this current study, including participants with POS or PGTC. Data for this outcome measure have been reported in relationship with different ranges of Cav, ss of Perampanel as "number of observations" those were seizure free for up to 3 visits. The reason for using number of observations for analysis of this outcome measure was because data were available as up to 3 visits per participant and not necessarily that the participant was seizure-free on all three visits.
Time Frame: Baseline up to Week 23
Population: as for outcome 5
Measure: Count of Units; unit: Seizure free observations
Units Other Than Participants: Seizure free observations
Groups:
- Perampanel: POS: All participants with POS who received perampanel 0.5 mg/mL oral suspension (for participants with age <12 years) or tablets (for participants with age >=12 years) titrated to a dose of up to 8 mg/day for up to 23 weeks in studies E2007-G000-304 (NCT00699972), E2007-G000-305 (NCT00699582), E2007-G000-306 (NCT00700310), E2007-J000-335 (NCT01618695) and this current study (E2007-G000-311).
Arm/Group | Perampanel: POS | Perampanel: PGTC Seizures
Number analyzed (Participants) | 1371 | 92
Number analyzed (Seizure free observations) | 3974 | 255
Seizure free observations
  >0 to <500 ng/mL: number analyzed (Seizure free observations) | 3189 | 127
  >0 to <500 ng/mL | 275 | 57
  500 to <1000 ng/mL: number analyzed (Seizure free observations) | 583 | 104
  500 to <1000 ng/mL | 103 | 67
  1000 to <1500 ng/mL: number analyzed (Seizure free observations) | 159 | 15
  1000 to <1500 ng/mL | 33 | 11
  1500 to 2000 ng/mL: number analyzed (Seizure free observations) | 33 | 6
  1500 to 2000 ng/mL | 7 | 4
  >2000 ng/mL: number analyzed (Seizure free observations) | 10 | 3
  >2000 ng/mL | 0 | 3

9. Secondary Outcome: Model Predicted Change From Baseline in Total Aldenkamp-Baker Neuropsychological Assessment Schedule (ABNAS) Score During Core Phase of This Study: Assessment Based on Relationship With Plasma Levels of Perampanel
Description: The ABNAS assessment measured 5 aspects of cognitive function such as fatigue, memory, concentration, motor speed, and reading. The assessment was a measure of participant-perceived cognitive effects of AEDs. This instrument was aimed at assessing participant perceived drug-related cognitive impairment. Total score ranged from 0-72. Higher scores indicate a worsening of these cognitive functions. Analysis for this outcome measure was planned to be performed via Pharmacokinetic/Pharmacodynamic (PK/PD) modelling only if a graphical relationship between perampanel exposure and change from baseline in ABNAS could be discerned.
Time Frame: Baseline up to Week 23
Population: All participants who received perampanel who have seizure frequency, cognition, or AE data with documented dosing history. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 148
score on a scale | NA (NA) — No discernible graphical relationship between plasma level of perampanel and change from baseline in ABNAS score was observed to warrant further PK/PD modelling and to summarize the data.

10. Secondary Outcome: Model Predicted Change From Baseline in Total Child Behavior Check List (CBCL) Score (Participants Aged 4 to 5 Years) During Core Phase of This Study: Assessment Based on Relationship With Plasma Levels of Perampanel
Description: The CBCL for participants with age 4 to 5 years is a questionnaire to assess behavioral and emotional problems in children as reported by the primary caregiver for the following domains activities: emotionally reactive, anxious/depressed, withdrawn, somatic complaints, internalizing, attention problems, aggressive behavior, externalizing, sleep problems. CBCL total score for participants with age 4 to 5 years ranged from 0 to 200, was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior. Analysis for this outcome measure was planned to be performed via PK/PD modelling only if a graphical relationship between perampanel exposure and change from baseline in CBCL score (participants aged 4 to 5 years) could be discerned.
Time Frame: Baseline up to Week 23
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 19
score on a scale | NA (NA) — No discernible graphical relationship between plasma level of perampanel and change from baseline in CBCL score (Participants Aged 4 to 5 Years) was observed to warrant further PK/PD modelling and to summarize the data.

11. Secondary Outcome: Model Predicted Change From Baseline in Total Child Behavior Check List (CBCL) Score (Participants Aged Greater Than [>] 5 to <12 Years) During Core Phase of This Study: Assessment Based on Relationship With Plasma Levels of Perampanel
Description: The CBCL for participants with age >5 to <12 years is a questionnaire to assess behavioral and emotional problems in children as reported by the primary caregiver for the following domains activities: activity, social, school, total competence, anxious/depressed, withdrawn/depressed, somatic complaints, internalizing, rule-breaking behavior, aggressive behavior, externalizing, social problems, thought problems, attention problems. CBCL total score for participants with age >5 to <12 years ranged from 0 to 240, was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior. Analysis for this outcome measure was planned to be performed via PK/PD modelling only if a graphical relationship between perampanel exposure and change from baseline in CBCL score (participants aged >5 to <12 years) could be discerned.
Time Frame: Baseline up to Week 23
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 115
score on a scale | NA (NA) — No discernible graphical relationship between plasma level of perampanel and change from baseline in CBCL Score (Participants Aged >5 to <12 Years) was observed to warrant further PK/PD modelling and to summarize the data.

12. Secondary Outcome: Model Predicted Change From Baseline in Total Time to Complete LGPT Score for Dominant Hand in Core Phase of This Study for All Participants Aged 4 to <12 Years: Assessment Based on Relationship With Plasma Levels of Perampanell
Description: The Lafayette Grooved Pegboard Test (LGPT) measures visuomotor skills. This test is a manipulative dexterity test that consist of a metal matrix of 25 holes with randomly positioned slots. Participants require to insert 10 grooved pegs into the holes. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task is timed and the scores are the time taken for the participant to complete all 10 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds are recorded for the time. An increase in score (longer time) indicate worsening of visuomotor skills. Analysis for this outcome measure was planned to be performed via PK/PD modelling only if a graphical relationship between perampanel exposure and change from baseline in Total Time to Complete LGPT Score for Dominant Hand could be discerned.
Time Frame: Baseline up to Week 23
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 117
seconds | NA (NA) — No discernible graphical relationship between plasma level of perampanel and change from baseline in LGPT Score for Dominant Hand was observed to warrant further PK/PD modelling and to summarize the data.

13. Secondary Outcome: Model Predicted Change From Baseline in Total Time to Complete LGPT Score for Non-dominant Hand in Core Phase of This Study for All Participants Aged 4 to <12 Years: Assessment Based on Relationship With Plasma Levels of Perampanel
Description: The Lafayette Grooved Pegboard Test (LGPT) measures visuomotor skills. This test is a manipulative dexterity test that consist of a metal matrix of 25 holes with randomly positioned slots. Participants require to insert 10 grooved pegs into the holes. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task is timed and the scores are the time taken for the participant to complete all 10 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds are recorded for the time. An increase in score (longer time) indicate worsening of visuomotor skills. Analysis for this outcome measure was planned to be performed via PK/PD modelling only if a graphical relationship between perampanel exposure and change from baseline in Total Time to Complete LGPT Score for Non-dominant Hand could be discerned.
Time Frame: Baseline up to Week 23
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 113
seconds | NA (NA) — No discernible graphical relationship between plasma level of perampanel and change from baseline in LGPT Score for Non-dominant Hand was observed to warrant further PK/PD modelling and to summarize the data.

14. Secondary Outcome: Percentage of Participants With Most Frequent Treatment Emergent Adverse Events (AEs) for Total Group of Participants That Were Considered Related to Perampanel- Core Phase of This Study
Time Frame: Baseline up to 23 weeks
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 180
percentage of participants
  Irritability/Aggression/Agitation | 12.8
  Nasopharyngitis | 14.7
  Influenza | 6.4
  Pyrexia | 9.0
  Somnolence | 13.5

15. Secondary Outcome: Change From Baseline in Aldenkamp-Baker Neuropsychological Assessment Schedule (ABNAS) Score as Per Seizure Type at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: The ABNAS assessment measured 5 aspects of cognitive function such as fatigue, memory, concentration, motor speed, and reading. The assessment was a measure of participant-perceived cognitive effects of AEDs. This instrument was aimed at assessing participant perceived drug-related cognitive impairment. Total score ranged from 0-72. Higher scores indicate a worsening of these cognitive functions.
Time Frame: Baseline, Week 23, Week 52
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure and number analyzed 'n' signifies participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Perampanel 0.5 mg/mL: POS: Core Phase: Participants with partial onset-seizures (POS) received perampanel 0.5 milligrams per milliliter (mg/mL) oral suspension titrated beyond 8 milligram per day (mg/day) up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any enzyme-inducing antiepileptic drug [EIAED]), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel once daily at optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed Core Phase, entered Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
- Perampanel 0.5 mg/mL: PGTC Seizures: Core Phase: Participants with primary generalized tonic clonic (PGTC) seizures received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any other EIAED), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel oral suspension once daily at the optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed the Core Phase, entered the Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 140 | 30
score on a scale
  Baseline | 17.7 (18.96) | 28.6 (21.01)
  Change from Baseline at Week 23: number analyzed (Participants) | 107 | 19
  Change from Baseline at Week 23 | -1.2 (12.77) | 3.3 (12.42)
  Change from Baseline at Week 52: number analyzed (Participants) | 95 | 17
  Change from Baseline at Week 52 | -3.9 (16.91) | -0.2 (14.67)

16. Secondary Outcome: Change From Baseline in Total Child Behavior Check List (CBCL) Score (Age Group 1.5 to 5 Years) as Per Seizure Type at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: The CBCL for participants (age group 1.5 to 5 years) is a questionnaire to assess behavioral and emotional problems in children as reported by the primary caregiver for the following domains activities: emotionally reactive, anxious/depressed, withdrawn, somatic complaints, internalizing, attention problems, aggressive behavior, externalizing, sleep problems. CBCL total score for participants (age group 1.5 to 5 years) ranged from 0 to 200, was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 24 | 2
score on a scale
  Baseline | 35.0 (28.30) | 54.0 (21.21)
  Change from Baseline at Week 23: number analyzed (Participants) | 15 | 1
  Change from Baseline at Week 23 | -0.3 (14.71) | -13.0 (NA) — Standard deviation could not be calculated because only one participants was available for analysis.
  Change from Baseline at Week 52: number analyzed (Participants) | 16 | 1
  Change from Baseline at Week 52 | -5.7 (14.36) | -11.0 (NA) — Standard deviation could not be calculated because only one participants was available for analysis.

17. Secondary Outcome: Change From Baseline in Total Child Behavior Check List (CBCL) Score (Age Group 6 to 18 Years) as Per Seizure Type at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: The CBCL for participants (age group 6 to 18 years) is a questionnaire to assess behavioral and emotional problems in children as reported by the primary caregiver for the following domains activities: activity, social, school, total competence, anxious/depressed, withdrawn/depressed, somatic complaints, internalizing, rule-breaking behavior, aggressive behavior, externalizing, social problems, thought problems, attention problems. CBCL total score for participants (age group 6 to 18 years) ranged from 0 to 240, was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 123 | 28
score on a scale
  Baseline | 33.3 (22.66) | 44.6 (26.16)
  Change from Baseline at Week 23: number analyzed (Participants) | 96 | 18
  Change from Baseline at Week 23 | -0.6 (12.26) | -2.2 (22.84)
  Change from Baseline at Week 52: number analyzed (Participants) | 86 | 16
  Change from Baseline at Week 52 | -1.7 (14.51) | -0.7 (16.36)

18. Secondary Outcome: Change From Baseline in Time to Complete Lafayette Grooved Pegboard Test (LGPT) Scores for 8 Years and Under as Per Seizure Type at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: The LGPT test measured visuomotor skills. This test was a manipulative dexterity test that consisted of a metal matrix of 25 holes with randomly positioned slots. The participant was required to insert 10 grooved pegs into the holes. The task was completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task was timed and the scores were the time taken for the participant to complete all 10 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds were recorded for the time. An increase in score (longer time) indicated worsening of visuomotor skills. The time to complete test is presented as mean seconds plus/minus (+/-) SD.
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 51 | 10
seconds
  Dominant Hand: Baseline | 196.4 (113.12) | 155.0 (108.10)
  Dominant Hand: Change from Baseline at Week 23: number analyzed (Participants) | 36 | 3
  Dominant Hand: Change from Baseline at Week 23 | 12.8 (49.37) | -4.3 (3.79)
  Dominant Hand: Change from Baseline at Week 52: number analyzed (Participants) | 28 | 5
  Dominant Hand: Change from Baseline at Week 52 | 3.9 (50.50) | 13.4 (33.72)
  Non Dominant Hand: Baseline: number analyzed (Participants) | 50 | 9
  Non Dominant Hand: Baseline | 224.3 (108.19) | 169.6 (106.49)
  Non Dominant Hand: Change from Baseline at Week 23: number analyzed (Participants) | 36 | 3
  Non Dominant Hand: Change from Baseline at Week 23 | 3.3 (39.59) | -4.3 (14.98)
  Non Dominant Hand: Change from Baseline at Week 52: number analyzed (Participants) | 29 | 5
  Non Dominant Hand: Change from Baseline at Week 52 | 2.6 (46.88) | 3.4 (29.35)

19. Secondary Outcome: Change From Baseline in Time to Complete Lafayette Grooved Pegboard Test (LGPT) Scores Over 8 Years as Per Seizure Type at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: The LGPT test measured visuomotor skills. This test was a manipulative dexterity test that consisted of a metal matrix of 25 holes with randomly positioned slots. The participant was required to insert 25 grooved pegs into the holes. The task was completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task was timed and the scores were the time taken for the participant to complete all 25 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds were recorded for the time. An increase in score (longer time) indicated worsening of visuomotor skills. The time to complete test is presented as mean seconds +/- SD.
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 63 | 11
seconds
  Dominant Hand: Baseline | 189.8 (103.58) | 150.7 (99.68)
  Dominant Hand: Change from Baseline at Week 23: number analyzed (Participants) | 50 | 9
  Dominant Hand: Change from Baseline at Week 23 | 0.1 (21.77) | -11.8 (35.05)
  Dominant Hand: Change from Baseline at Week 52: number analyzed (Participants) | 44 | 7
  Dominant Hand: Change from Baseline at Week 52 | 3.0 (21.24) | -15.4 (30.43)
  Non Dominant Hand: Baseline: number analyzed (Participants) | 61 | 10
  Non Dominant Hand: Baseline | 197.4 (100.01) | 159.9 (84.66)
  Non Dominant Hand: Change from Baseline at Week 23: number analyzed (Participants) | 49 | 8
  Non Dominant Hand: Change from Baseline at Week 23 | 7.8 (36.03) | -7.0 (21.98)
  Non Dominant Hand: Change from Baseline at Week 52: number analyzed (Participants) | 42 | 6
  Non Dominant Hand: Change from Baseline at Week 52 | 2.7 (23.75) | -28.7 (36.15)

20. Secondary Outcome: Change From Baseline in Height (a Growth and Development Parameter) at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 149 | 29
centimeter (cm)
  Baseline | 126.65 (14.293) | 131.08 (13.311)
  Change from Baseline Week 23: number analyzed (Participants) | 114 | 18
  Change from Baseline Week 23 | 2.57 (1.926) | 1.84 (1.111)
  Change from Baseline Week 52: number analyzed (Participants) | 104 | 17
  Change from Baseline Week 52 | 5.97 (2.580) | 5.82 (2.544)

21. Secondary Outcome: Change From Baseline in Weight (a Growth and Development Parameter) at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Time Frame: Baseline, Week 23, Week 52
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Here number analyzed 'n' signifies participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 149 | 31
kilogram (kg)
  Baseline | 28.09 (10.649) | 30.43 (11.299)
  Change from Baseline at Week 23: number analyzed (Participants) | 117 | 21
  Change from Baseline at Week 23 | 1.86 (2.570) | 1.70 (3.149)
  Change from Baseline at Week 52: number analyzed (Participants) | 104 | 18
  Change from Baseline at Week 52 | 3.75 (4.421) | 3.74 (4.204)

22. Secondary Outcome: Change From Baseline in Thyrotropin Value (a Growth and Development Parameter) at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Description: Thyrotropin level was measured in milli-international units per liter (mIU/L).
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 146 | 30
mIU/L
  Baseline | 2.682 (1.5897) | 3.080 (2.2919)
  Change from Baseline at Week 23: number analyzed (Participants) | 104 | 17
  Change from Baseline at Week 23 | 0.141 (1.0523) | -0.519 (1.4828)
  Change from Baseline at Week 52: number analyzed (Participants) | 97 | 17
  Change from Baseline at Week 52 | 0.112 (1.2559) | -0.632 (1.5632)

23. Secondary Outcome: Change From Baseline in Thyroxine, Free and Triiodothyronine, Free Values (Growth and Development Parameters) at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 146 | 30
picomoles per liter (pmol/L)
  Thyroxine, free: Baseline | 15.29 (3.993) | 15.37 (2.160)
  Thyroxine, free: Change at Week 23: number analyzed (Participants) | 103 | 17
  Thyroxine, free: Change at Week 23 | -0.07 (4.107) | -0.38 (2.088)
  Thyroxine, free: Change at Week 52: number analyzed (Participants) | 96 | 17
  Thyroxine, free: Change at Week 52 | 0.10 (3.868) | 0.08 (2.968)
  Triiodothyronine, free: Baseline | 5.96 (1.061) | 6.10 (0.812)
  Triiodothyronine, free: Change at Week 23: number analyzed (Participants) | 105 | 18
  Triiodothyronine, free: Change at Week 23 | 0.06 (0.915) | -0.16 (0.699)
  Triiodothyronine, free: Change at Week 52: number analyzed (Participants) | 96 | 17
  Triiodothyronine, free: Change at Week 52 | 0.04 (0.987) | -0.04 (1.107)

24. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor-1 (IGF-1) Values (a Growth and Development Parameter) at Week 23 (Core Phase) and at Week 52 (Extension Phase A) of This Study
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 144 | 31
nanomoles per liter (nmol/L)
  Baseline | 24.2 (14.83) | 25.9 (13.91)
  Change from Baseline Week 23: number analyzed (Participants) | 107 | 18
  Change from Baseline Week 23 | 1.6 (8.96) | 0.6 (7.25)
  Change from Baseline Week 52: number analyzed (Participants) | 96 | 16
  Change from Baseline Week 52 | 6.5 (9.01) | 5.1 (8.02)

25. Secondary Outcome: Percentage of Participants With Change From Baseline in Markedly Abnormal Encephalogram (EEG) Parameter Values During Awake and Sleep State for Total Group of Participant: Core Phase and Extension Phase A of This Study
Time Frame: Baseline up to 52 weeks
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 180
percentage of participants | 0

26. Secondary Outcome: Number of Encephalogram (EEG) Abnormalities During Awake and Sleep State for Total Group of Participant: Core Phase and Extension Phase A of This Study
Time Frame: Baseline up to 52 weeks
Population: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: EEG abnormality
Arm/Group | Perampanel 0.5 mg/mL: All Participants
Number analyzed (Participants) | 180
EEG abnormality | 0

27. Secondary Outcome: Percentage of Participants With Any Treatment-emergent Reports of Suicidal Ideation and Behavior Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS)- Core Phase and Extension Phase A of This Study
Description: C-SSRS: interview-based instrument to systematically assess suicidal ideation (SI) and behavior, to assess whether participant experienced any of following: completed suicide, suicide attempt (response of "yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior ("yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active SI with methods without intent to act or some intent to act, without or with specific plan and intent), any self-injurious behavior with no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior").Here, percentage of participants with >=1 positive behavior, participants with >=1 positive ideations; suicidality were reported.An assessment of SI and behavior with C-SSRS performed for participants >=6 years at time of consent.
Time Frame: Up to 52 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 122 | 27
percentage of participants
  Participants with >=1 Positive Behavior | 0.8 | 0
  Participants with >= Positive Ideations | 1.6 | 7.4
  Suicidality | 1.6 | 7.4

28. Secondary Outcome: Percentage of Participants With Shift From Baseline in Suicidal Ideation and Behaviors Assessed Using C-SSRS Scores to Extension Phase A (Week 52) of This Study
Description: The C-SSRS: interview-based instrument to systematically assess suicidal ideation (SI) and suicidal behavior, to assess whether participant experienced any of the following: completed suicide, suicide attempt (response of "yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior ("yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active SI with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any self-injurious behavior with no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). "w/" refers to "with", "W" refers to "Week" and "&" refers to "and".
Time Frame: Up to 52 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 122 | 27
percentage of participants
  No Ideation (Baseline) to No Ideation(Week 52) | 96.6 | 88.9
  Wish to be Dead(Baseline) to No ideation(Week 52) | 0.9 | 3.7
  Active w/ Method(Baseline) to No Ideation(Week 52) | 0.9 | 0
  No Ideation(Baseline)to Active Nonspecific(Week52) | 0 | 3.7
  No Ideation(Baseline) to Active w/ Method(Week 52 | 0.9 | 3.7
  No Ideation(Baseline)to Active w/ Intent&Plan(W52) | 0.9 | 0

29. Secondary Outcome: Median Percent Change in Seizure Frequency Per 28 Days During the Treatment Phase Relative to the Pretreatment Phase (Baseline)- Core Phase and Extension Phase A of This Study
Description: Seizure frequency was based on number of seizures per 28 days, calculated as number of seizures over entire time interval divided by number of days in interval and multiplied by 28. Total POS: sum of all POS including simple partial seizures without motor signs, simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with secondary generalization (SG). Data for this measure has been reported for 13 week time periods as per age groups.
Time Frame: Baseline, Weeks 1-13, Weeks 14-26, Weeks 27-39, Weeks 40-52
Population: Full Analysis Set (FAS) included participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Here overall number of participants analyzed 'N' signifies participants who were evaluable for this outcome measure and number analyzed 'n' signifies participants who were evaluable for specified timepoints.
Measure: Median (Full Range); unit: percent change
Groups:
- Perampanel 0.5 mg/mL: 4 to <7 Years: Core Phase: Participants of age 4 to <7 years with POS or PGTC seizures received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any EIAED), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel once daily at optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed Core Phase, entered Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
- Perampanel 0.5 mg/mL: 7 to <12 Years: Core Phase: Participants of age 7 to <12 years with POS or PGTC seizures received perampanel 0.5 mg/mL oral suspension titrated beyond 8 mg/day up to 12 mg/day, if 8 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are not taking any other EIAED), or titrated beyond 12 mg/day up to 16 mg/day, if 12 mg/day was tolerable and were deemed likely to be benefitted by higher dose (for participants who are taking any EIAED). Dose titration- up to 11 weeks to identify each participant's optimum dose. Participants then continued to take perampanel oral suspension once daily at the optimal dose level as a maintenance dose for up to 12 weeks. Extension Phase A: Participants who completed the Core Phase, entered the Extension Phase A, and continued with their optimal perampanel dose from Core Phase for up to 29 weeks. Total duration of treatment for Core Phase and Extension Phase A was up to 52 weeks.
Arm/Group | Perampanel 0.5 mg/mL: 4 to <7 Years | Perampanel 0.5 mg/mL: 7 to <12 Years
Number analyzed (Participants) | 40 | 108
percent change
  POS Seizures:Weeks 1-13 | -47.99 [-100.0 to 79.1] | -40.97 [-100.0 to 549.0]
  POS Seizures:Weeks 14-26: number analyzed (Participants) | 39 | 91
  POS Seizures:Weeks 14-26 | -38.93 [-100.0 to 175.0] | -50.77 [-100.0 to 360.5]
  POS Seizures:Weeks 27-39: number analyzed (Participants) | 32 | 82
  POS Seizures:Weeks 27-39 | -52.53 [-100.0 to 344.2] | -67.30 [-100.0 to 387.9]
  POS Seizures:Weeks 40-52: number analyzed (Participants) | 31 | 77
  POS Seizures:Weeks 40-52 | -58.92 [-100.0 to 482.7] | -70.33 [-100.0 to 436.3]
  PGTC Seizures:Weeks 1-13: number analyzed (Participants) | 3 | 19
  PGTC Seizures:Weeks 1-13 | -100.00 [-100.0 to 2115.9] | -70.33 [-100.0 to 6783.5]
  PGTC Seizures:Weeks 14-26: number analyzed (Participants) | 3 | 15
  PGTC Seizures:Weeks 14-26 | -100.00 [-100.0 to -7.7] | -70.70 [-100.0 to 879.1]
  PGTC Seizures:Weeks 27-39: number analyzed (Participants) | 2 | 13
  PGTC Seizures:Weeks 27-39 | -80.77 [-100.0 to -61.5] | -65.43 [-100.0 to 315.4]
  PGTC Seizures:Weeks 40-52: number analyzed (Participants) | 2 | 11
  PGTC Seizures:Weeks 40-52 | -100.00 [-100.0 to -100.0] | -96.54 [-100.0 to 658.4]

30. Secondary Outcome: Percentage of Participants Based on 25% Responder Rate- Core Phase and Extension Phase A of This Study
Description: A 25% responder was a participant who experienced a 25% or greater reduction in seizure frequency per 28 days from baseline. Total POS: sum of all POS including simple partial seizures without motor signs, simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with SG. Data for this outcome measure has been reported for 13 week time periods as per age groups.
Time Frame: Baseline, Weeks 1-13, Weeks 14-26, Weeks 27-39, Weeks 40-52
Population: FAS included participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: 4 to <7 Years | Perampanel 0.5 mg/mL: 7 to <12 Years
Number analyzed (Participants) | 46 | 134
percentage of participants
  Total POS Seizures: Weeks 1-13 | 67.5 | 61.1
  Total POS Seizures: Weeks 14-26 | 57.9 | 71.4
  Total POS Seizures: Weeks 27-39 | 71.9 | 78.0
  Total POS Seizures: Weeks 40-52 | 71.0 | 81.8
  PGTC Seizures: Weeks 1-13 | 66.7 | 73.7
  PGTC Seizures: Weeks 14-26 | 66.7 | 73.3
  PGTC Seizures: Weeks 27-39 | 100.0 | 69.2
  PGTC Seizures: Weeks 40-52 | 100.0 | 63.6

31. Secondary Outcome: Percentage of Participants Based on 50% Responder Rate- Core Phase and Extension Phase A of This Study
Description: A 50% responder was a participant who experienced a 50% or greater reduction in seizure frequency per 28 days from baseline. Total POS: sum of all POS including simple partial seizures without motor signs, simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with SG. Data for this outcome measure has been reported for 13 week time periods as per age groups.
Time Frame: Baseline, Weeks 1-13, Weeks 14-26, Weeks 27-39, Weeks 40-52
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: 4 to <7 Years | Perampanel 0.5 mg/mL: 7 to <12 Years
Number analyzed (Participants) | 46 | 134
percentage of participants
  Total POS Seizures: Weeks 1-13 | 47.5 | 45.4
  Total POS Seizures: Weeks 14-26 | 44.7 | 50.5
  Total POS Seizures: Weeks 27-39 | 53.1 | 65.9
  Total POS Seizures: Weeks 40-52 | 61.3 | 62.3
  PGTC Seizures: Weeks 1-13 | 66.7 | 57.9
  PGTC Seizures: Weeks 14-26 | 66.7 | 60.0
  PGTC Seizures: Weeks 27-39 | 100.0 | 61.5
  PGTC Seizures: Weeks 40-52 | 100.0 | 54.5

32. Secondary Outcome: Percentage of Participants Based on 75% Responder Rate- Core Phase and Extension Phase A of This Study
Description: A 75% responder was a participant who experienced a 75% or greater reduction in seizure frequency per 28 days from baseline. Total POS: sum of all POS including simple partial seizures without motor signs, simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with SG. Data for this outcome measure has been reported for 13 week time periods as per age groups.
Time Frame: Baseline, Weeks 1-13, Weeks 14-26, Weeks 27-39, Weeks 40-52
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: 4 to <7 Years | Perampanel 0.5 mg/mL: 7 to <12 Years
Number analyzed (Participants) | 46 | 134
percentage of participants
  Total POS Seizures: Weeks 1-13 | 17.5 | 25.0
  Total POS Seizures: Weeks 14-26 | 18.4 | 34.1
  Total POS Seizures: Weeks 27-39 | 31.3 | 46.3
  Total POS Seizures: Weeks 40-52 | 38.7 | 41.6
  PGTC Seizures: Weeks 1-13 | 66.7 | 47.4
  PGTC Seizures: Weeks 14-26 | 66.7 | 46.7
  PGTC Seizures: Weeks 27-39 | 50.0 | 46.2
  PGTC Seizures: Weeks 40-52 | 100.0 | 54.5

33. Secondary Outcome: Percentage of Participants Who Were Seizure-free- Core Phase and Extension Phase A of This Study
Description: Participants were considered seizure free if participants completed a 13-week time period and were seizure-free for that entire time period. Total POS: sum of all POS including simple partial seizures without motor signs, simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with SG. Data for this outcome measure has been reported for 13 week time periods as per age groups.
Time Frame: Weeks 1-13, Weeks 14-26, Weeks 27-39, Weeks 40-52
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: 4 to <7 Years | Perampanel 0.5 mg/mL: 7 to <12 Years
Number analyzed (Participants) | 46 | 134
percentage of participants
  Total POS Seizures: Weeks 1-13 | 7.9 | 9.9
  Total POS Seizures: Weeks 14-26 | 9.4 | 15.9
  Total POS Seizures: Weeks 27-39 | 12.9 | 24.7
  Total POS Seizures: Weeks 40-52 | 15.0 | 20.8
  PGTC Seizures: Weeks 1-13 | 66.7 | 40.0
  PGTC Seizures: Weeks 14-26 | 50.0 | 46.2
  PGTC Seizures: Weeks 27-39 | 50.0 | 45.5
  PGTC Seizures: Weeks 40-52 | 100.0 | 57.1

34. Secondary Outcome: Percentage of Participants With Clinical Global Impression of Change Scores (CGIC)- Core Phase and Extension Phase A of This Study
Description: Assessment of disease severity utilized the CGIC scale at end of treatment to evaluate participant's change in disease status from baseline. The CGIC is a 7-point scale that measures a physician's global impression of a participant's clinical condition. Scale ranged from 1 to 7 with lower score indicated improvement (1=very much improved, 2=much improved, 3=minimally improved), higher score indicated worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicated no change.
Time Frame: Baseline, Week 23, Week 52
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 0.5 mg/mL: POS | Perampanel 0.5 mg/mL: PGTC Seizures
Number analyzed (Participants) | 149 | 31
percentage of participants
  Week 23: Very much improved | 11.5 | 8.7
  Week 23: Much improved | 31.1 | 26.1
  Week 23: Minimally improved | 38.5 | 26.1
  Week 23: No change | 14.8 | 26.1
  Week 23: Minimally worse | 3.3 | 13.0
  Week 23: Much worse | 0.8 | 0
  Week 52: Very much improved | 14.4 | 5.9
  Week 52: Much improved | 39.4 | 41.2
  Week 52: Minimally improved | 35.6 | 29.4
  Week 52: No change | 7.7 | 17.6
  Week 52: Minimally worse | 1.9 | 5.9
  Week 52: Much worse | 1.0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to approximately 5 years
Description: SAS included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Arm/Group | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures | Extension B: Perampanel 0.5 mg/mL: POS | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures
All-Cause Mortality (participants affected / at risk) | 1/149 | 0/31 | 0/41 | 0/1
Serious Adverse Events (participants affected / at risk) | 29/149 | 7/31 | 8/41 | 0/1
Other Adverse Events (participants affected / at risk) | 135/149 | 25/31 | 34/41 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS (N=149) | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures (N=31) | Extension B: Perampanel 0.5 mg/mL: POS (N=41) | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures (N=1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (7) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (7) | 0 (0) | 5 (6) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rasmussen encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Study + Extension Part A: Perampanel 0.5 mg/mL: POS (N=149) | Core Study + Extension Part A: Perampanel 0.5 mg/mL: PGTC Seizures (N=31) | Extension B: Perampanel 0.5 mg/mL: POS (N=41) | Extension B: Perampanel 0.5 mg/mL: PGTC Seizures (N=1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Corneal disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (5) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 3 (5) | 3 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 20 (23) | 5 (6) | 5 (13) | 0 (0)
Rubber sensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 10 (11) | 0 (0) | 4 (6) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 11 (14) | 2 (2) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 20 (23) | 0 (0) | 6 (6) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 40 (73) | 3 (4) | 14 (25) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 6 (8) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (5) | 3 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 3 (3) | 3 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mallet finger (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 6 (10) | 2 (2) | 0 (0) | 0 (0)
Atonic seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 4 (8) | 3 (3) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 19 (24) | 5 (8) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyslexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysstasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Persistent postural-perceptual dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Postictal state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 5 (6) | 2 (3) | 0 (0) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 6 (9) | 3 (4) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 43 (49) | 5 (9) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 15 (22) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 7 (11) | 2 (2) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Defiant behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphemia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 1 (3) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 19 (20) | 5 (5) | 1 (1) | 0 (0)
Learning disability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Negativism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (7) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (13) | 1 (1) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Crying (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (11) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 25 (39) | 4 (6) | 4 (4) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (5) | 1 (1) | 4 (5) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (18) | 5 (7) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ranula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Screaming (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perianal streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periosteal haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hippocampal sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Simple partial seizures (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Distractibility (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Precocious puberty (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lagophthalmos (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema infectiosum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site erosion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blast cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT02849626/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02849626/SAP_001.pdf